CLINICAL TRIAL: NCT00630604
Title: Quantitative Evaluation by Ultrasonography for Severity of Knee Osteoarthritis
Brief Title: Quantitative Ultrasonography (US) Evaluation on Femoral Condyle Cartilage
Acronym: US
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Chia-Ling Lee, Kaohsiung Medical University Hospital
Other Study IDs: NSC 94-2314-B-037-020; NSC 94-2314-B-037-020
Record Dates: First submitted 2008-02-22; First posted 2008-03-07 (Estimated); Last update posted 2008-03-07 (Estimated); Status verified 2008-02

CONDITIONS: Osteoarthritis
Keywords: ultrasonography; knee; early degeneration; cartilage
MeSH Terms: conditions — Osteoarthritis

SUMMARY:
The purpose of this study is to investigate the feasibility of using quantitative ultrasonography (US) evaluation to determine the severity of osteoarthritic femoral condyle cartilage erosion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with knee OA who were going to receive total knee arthroplasty

Exclusion Criteria:

* Patients with inflammatory arthritis (e.g. rheumatic arthritis) and infectious disease (e.g. hepatitis B)

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with knee OA who were going to receive total knee arthroplasty
Sampling Method: Probability Sample

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling Lee, MS, Principal Investigator — MD